CLINICAL TRIAL: NCT02515656
Title: Assessment of the Efficacy of POLYGYNAX® in the Empirical Treatment of Infectious Vaginitis International, Multicentre, Randomised, Double-blind, Parallel Group Study, Comparative Versus Miconazole
Brief Title: Assessment of the Efficacy of POLYGYNAX® in the Empirical Treatment of Infectious Vaginitis
Acronym: PRISM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoire Innotech International (Industry)
Collaborators: International Clinical Trials Association (Other); Venn Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGX 401-11; 2014-001759-22 (EudraCT Number)
Record Dates: First submitted 2015-07-29; First posted 2015-08-05 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-08

CONDITIONS: Vaginitis
MeSH Terms: conditions — Vaginitis | interventions — acetarsol, dimethicone, neomycin, nystatin, polymyxin drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- POLYGYNAX® (Experimental): Name : POLYGYNAX® Active components : nystatin 100 000 IU + neomycin sulphate 35 000 IU + polymyxin B sulphate 35 000 IU Dosage : 1 capsule intravaginally per day (administered at bedtime lying down) 12 vaginal soft capsules
  Interventions: Drug: POLYGYNAX®
- miconazole + placebo (Active Comparator): Name : GYNODAKTARIN® Active components : miconazole nitrate 400 mg Dosage : 1 capsule intravaginally per day (administered at bedtime, lying down) 3 vaginal soft capsules followed by 9 placebo vaginal soft capsules
  Interventions: Drug: GYNODAKTARIN®; Drug: Placebo

INTERVENTIONS:
Drug: POLYGYNAX®
  Arms: POLYGYNAX®
Drug: GYNODAKTARIN®
  Arms: miconazole + placebo
Drug: Placebo
  Arms: miconazole + placebo

SUMMARY:
POLYGYNAX® is a broad spectrum combination of nystatin, neomycin and polymixin B indicated for the local treatment of vaginitis due to sensitive germs and treatment of non specific vaginitis of adults. POLYGYNAX® has been marketed in France since 1969.

Nevertheless, despite the well established use of POLYGYNAX®, there is no clinical study supporting the interest of the combination of antifungal and antibiotics agents versus antifungal agent alone.

The aim of this project is to demonstrate that POLYGYNAX® is more effective than miconazole in the treatment of women experiencing symptoms of infectious vaginitis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an abnormal vaginal discharge associated with one (or more) functional vaginal complaints: vaginal burning and/or vaginal pain and/or vaginal irritation clinically evoking an infectious vaginitis:

  * bacterial vaginitis
  * non-specific vaginitis (atypical symptoms)
  * mixed vaginitis (i.e. suprainfected fungal vaginitis) and able to receive an empirical local treatment

Exclusion Criteria:

1. Recurrent patient; i.e. a patient who has had at least 4 episodes of infectious vaginitis in the 12 months prior to inclusion
2. Vaginal infection justifying systemic therapy
3. History of atrophic vaginitis or suspected atrophic vaginitis at inclusion
4. Patient presenting with signs of genital herpes or signs of non-infectious vulvar pathology (vulvodynia, psoriasis, eczema, lichen sclerosus, lichen planus, contact dermatitis, candida intertrigo, vulval intraepithelial neoplasia (VIN))
5. Patient with current Sexually Transmitted Infection (STI) and/or patients with clinical suspicion of STI
6. Disease or concomitant treatment that could cause decreased immunity (i.e. diabetes mellitus, corticosteroids treatments)
7. Systemic anti-infective treatment (antibiotic, antifungal) within two weeks prior to inclusion
8. Patient menstruating or patient with menometrorrhagia due to hormonal imbalance at the time of inclusion
9. Pregnant or lactating women or delivery within last 1 month

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 661 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc BOHBOT, Dr, Principal Investigator — Institut Alfred Fournier
Locations (4):
- TURKOVA, Prague, Czechia
- PERCEVAL, Lyon, France
- MARICIC, Belgrade, Serbia
- GATOVA, Martin, Slovakia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 patients who signed an Informed Consent Form (ICF) were screen failed and were not randomized in the study.
Groups:
- POLYGYNAX®: Name : POLYGYNAX® Active components : nystatin 100 000 IU + neomycin sulphate 35 000 IU + polymyxin B sulphate 35 000 IU Dosage : 1 capsule intravaginally per day (administered at bedtime lying down) 12 vaginal soft capsules
  POLYGYNAX®
- Miconazole + Placebo: Name : GYNODAKTARIN® Active components : miconazole nitrate 400 mg Dosage : 1 capsule intravaginally per day (administered at bedtime, lying down) 3 vaginal soft capsules followed by 9 placebo vaginal soft capsules
  GYNODAKTARIN®
  Placebo
Period: Overall Study
Arm/Group | POLYGYNAX® | Miconazole + Placebo
Started | 326 | 332
Full Analysis Set (FAS) | 302 | 309
Per Protocol Set (PPS) | 277 | 275
Safety Population | 325 | 328
Completed | 270 | 261
Not Completed | 56 | 71

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | POLYGYNAX® | Miconazole + Placebo | Total
Number analyzed (Participants) | 302 | 309 | 611
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.70 (10.13) | 33.73 (10.07) | 34.21 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 302 | 309 | 611
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Treatment Efficacy Assessed by the Investigator After Thorough Gynaecological Examination and Patient's Interview at End of Treatment Visit
Description: * Success is defined by resolution (return to patient's usual gynaecological conditions, i.e. before the episode which warranted inclusion in the study) OR substantial improvement of clinical signs of infectious vaginitis (i.e. abnormal vaginal discharge), and/or vaginal symptoms (vaginal burning and/or vaginal pain, and/or vaginal irritation).
  * Failure is defined by persistence or worsening of symptoms and clinical signs or requirement of an alternative or specific treatment.
  Not considered as "Treatment Failure":
  * The need to initiate a specific treatment because of a Sexually Transmitted Infection (STI) (trichomoniasis; gonococcal and chlamydial infections) detected from the vaginal sample at Visit 1 / D1.
  * Patients presenting with only vulvar complaints not considered as related to infectious vaginitis.
Time Frame: 15 days after first treatment administration
Measure: Count of Participants; unit: Participants
Arm/Group | POLYGYNAX® | Miconazole + Placebo
Number analyzed (Participants) | 302 | 309
Participants
  Success | 275 | 268
  Failure | 27 | 41

2. Secondary Outcome: Change in Vaginal Discharge and in Each Associated Vaginal Clinical Symptoms Reported by the Patient in the Diary
Description: This outcome was evaluated using a Visual Analogue Scale (VAS) completed by the patient.
  The scale measured the level of each vaginal symptom experienced during the day (vaginal discharge, vaginal burning, vaginal pain and vaginal irritation).
  Scale ranges = 0 to 100 0=none symptom 100=maximum intensity of symptom Time points used in the calculation= D1 to D14
Time Frame: during 14 days after first treatment intake
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | POLYGYNAX® | Miconazole + Placebo
Number analyzed (Participants) | 302 | 309
mm
  Vaginal discharge absolute change | 31.43 [29.94 to 32.91] | 29.54 [28.07 to 31.01]
  Vaginal burning absolute change | 27.89 [26.66 to 29.12] | 27.03 [25.81 to 28.25]
  Vaginal pain absolute change | 16.93 [15.86 to 18.01] | 17.17 [16.10 to 18.24]
  Vaginal irritation absolute change | 29.37 [28.06 to 30.67] | 28.79 [27.51 to 30.08]
  Vaginal combined clinical symptoms score absolute | 28.96 [26.79 to 31.14] | 28.20 [26.04 to 30.35]

3. Secondary Outcome: Number of Patients With Change in Vaginal Discharge Assessed by the Investigator
Description: The vaginal discharge is assessed by the investigator by using a score:
  0=absent
  1. mild: insufficient for speculum collection
  2. moderate: sufficient for speculum collection
  3. abundant: visible at the introitus even before speculum introduction.
Time Frame: 15 days after first treatment administration
Measure: Count of Participants; unit: Participants
Arm/Group | POLYGYNAX® | Miconazole + Placebo
Number analyzed (Participants) | 300 | 307
Participants
  Leucorrhoea score change - Deterioration | 1 | 7
  Leucorrhoea score change - No change | 19 | 24
  Leucorrhoea score change - Improvement | 280 | 276

4. Secondary Outcome: Clinical Treatment Efficacy (Success/Failure) Assessed by the Investigator After Thorough Gynaecological Examination and Patient's Interview at End of Study Visit
Description: Success and Failure (same definition as the primary outcome measure)
Time Frame: 22 days after first treatment administration
Population: There were 5 and 6 missing values respectively in Polygynax and Miconazole + placebo arms.
Measure: Count of Participants; unit: Participants
Arm/Group | POLYGYNAX® | Miconazole + Placebo
Number analyzed (Participants) | 302 | 309
Participants
  Success: number analyzed (Participants) | 297 | 303
  Success | 252 | 250
  Failure: number analyzed (Participants) | 297 | 303
  Failure | 45 | 53

5. Secondary Outcome: Investigator's Global Satisfaction
Description: The investigator filled the satisfaction questionnaire during the end of treatment visit.
  Six ratings are available: Very Bad, Bad, Somewhat Bad, Somewhat Good, Good and Very Good.
Time Frame: 15 days after first administration
Measure: Count of Participants; unit: Participants
Arm/Group | POLYGYNAX® | Miconazole + Placebo
Number analyzed (Participants) | 300 | 307
Participants
  Very good - Good | 265 | 252
  Somewhat good - Somewhat bad | 25 | 40
  Bad - Very bad | 10 | 15

6. Secondary Outcome: Patient's Global Satisfaction
Description: The patient filled the satisfaction questionnaire on her patient's diary at home the eve of the End of Treatment Visit.
  Six ratings are available: Very Bad, Bad, Somewhat Bad, Somewhat Good, Good and Very Good.
Time Frame: 15 days after first administration
Population: There were 10 and 11 missing values respectively in Polygynax and Miconazole + placebo arms.
Measure: Count of Participants; unit: Participants
Arm/Group | POLYGYNAX® | Miconazole + Placebo
Number analyzed (Participants) | 292 | 298
Participants
  Very good - Good | 239 | 233
  Somewhat good - Somewhat bad | 50 | 63
  Bad - Very bad | 3 | 2

ADVERSE EVENTS:
Time Frame: 22 days
Arm/Group | POLYGYNAX® | Miconazole + Placebo
All-Cause Mortality (participants affected / at risk) | 0/325 | 0/328
Serious Adverse Events (participants affected / at risk) | 1/325 | 0/328
Other Adverse Events (participants affected / at risk) | 18/325 | 5/328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | POLYGYNAX® (N=325) | Miconazole + Placebo (N=328)
Patient pregnant exposed to study medications (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | POLYGYNAX® (N=325) | Miconazole + Placebo (N=328)
Headache (Nervous system disorders) | 18 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes